CLINICAL TRIAL: NCT07092319
Title: Impact of Delayed Cord Clamping and Minimally Invasive Surfactant Administration on Outcomes in Premature Infants With Neonatal Respiratory Distress Syndrome at Less Than 30 Weeks Gestation: A NICU Quality Improvement Study
Brief Title: Impact of Delayed Cord Clamping and Minimally Invasive Surfactant Administration on Outcomes in Premature Infants Less Than 30 Weeks Gestation
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024376
Record Dates: First submitted 2024-05-28; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: NRDS
Keywords: Delayed cord clamping; minimally invasive surfactant administration; preterm infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DCC+MISA group: Infants without contraindications to DCC, as determined by prenatal evaluation, receive immediate non-invasive respiratory support after birth. DCC is successfully performed for 60 seconds, followed by a diagnosis of NRDS. A therapeutic dose of pulmonary surfactant (PS) is administered via MISA within the first 2 hours after birth.
  Interventions: Procedure: deferred cord clamping
- ICC+tracheal intubation group: Umbilical cord clamping occurs within 20 seconds after birth. Infants are diagnosed with NRDS and receive a therapeutic dose of PS via tracheal intubation within the first 12 hours after birth.
- ICC+MISA group: Umbilical cord clamping is performed within 20 seconds after birth. Infants are diagnosed with NRDS and receive a therapeutic dose of PS via MISA within the first 2 hours after birth.

INTERVENTIONS:
Procedure: deferred cord clamping — DCC: deferred cord clamping successfully for 60 seconds;MISA: Surfactant administration by minimally invasive methods that allow for spontaneous breathing.
  Other Names: minimally invasive surfactant administration
  Groups: DCC+MISA group

SUMMARY:
Background:

Preventing early exposure to invasive mechanical ventilation in premature infants is crucial for reducing the incidence of bronchopulmonary dysplasia (BPD) and improving overall outcomes. Compared to immediate cord clamping (ICC) and tracheal intubation for pulmonary surfactant administration at birth, delayed cord clamping (DCC) combined with minimally invasive surfactant administration (MISA) has been shown to enhance early respiratory and circulatory stability in premature infants, thereby decreasing the need for invasive mechanical ventilation. The investigators hypothesize that for preterm infants under 30 weeks gestation diagnosed with respiratory distress syndrome (RDS), the combination of DCC and MISA will more effectively reduce the incidence of BPD.

Methods and Design:

The investigators will conduct a single-center ambispective cohort study to compare three treatment regimens in premature infants diagnosed with neonatal respiratory distress syndrome (NRDS) at less than 30 weeks gestation: Delayed cord clamping (DCC) combined with minimally invasive surfactant administration (MISA) (n=74); Immediate cord clamping (ICC) combined with tracheal intubation for pulmonary surfactant administration (n=222); Immediate cord clamping (ICC) combined with MISA (n=222). The study aims to evaluate the incidence of bronchopulmonary dysplasia (BPD), short-term treatment effects, safety, and long-term outcomes associated with each regimen, providing valuable evidence for clinical treatment decisions.

Discussion:

Current research indicates that both delayed cord clamping (DCC) and minimally invasive surfactant administration (MISA) positively impact the prognosis of very premature infants and help reduce the incidence of bronchopulmonary dysplasia (BPD). However, there is limited research on whether the combined use of DCC and MISA can further enhance survival rates and decrease BPD incidence in this vulnerable population.

The investigators NICU has gradually implemented MISA in respiratory management since 2017 and adopted cord management with DCC since 2023. This study retrospectively analyzes data from previous groups: those receiving immediate cord clamping (ICC) with MISA, and those receiving ICC with tracheal intubation. The investigators will compare this with prospective data from the DCC combined with MISA group to assess differences in BPD occurrence, other complications and overall outcomes.

Through this study, the investigators aim to determine whether the combination of DCC and MISA offers greater benefits in improving the prognosis of very premature infants, ultimately providing a stronger foundation for early respiratory and circulatory management strategies for infants born before 30 weeks.

DETAILED DESCRIPTION:
With the rapid advancement of neonatal intensive care technology, the survival rate of premature infants born at less than 30 weeks gestation continues to rise. However, the immaturity of various organ systems leads to a high incidence of complications, and long-term outcomes can often be less than optimistic[1]. Consequently, enhancing both short-term and long-term prognoses for these infants through quality improvement initiatives has become a prominent focus in recent clinical research.

Bronchopulmonary dysplasia (BPD) is a critical complication in very premature infants, significantly affecting their future survival, as well as their respiratory and neurological development. Preventing and reducing the incidence of BPD is crucial for improving the overall prognosis of these infants[2]. Ensuring postpartum respiratory and circulatory stability while minimizing exposure to early invasive mechanical ventilation is essential for preventing and reducing the incidence of BPD.

The management of respiratory and circulatory conditions in preterm infants begins with delayed umbilical cord clamping (DCC) in the delivery room. Compared to immediate cord clamping (ICC), DCC facilitates the transfer of blood from the placenta to the infant, enhancing the adaptability of vital organs such as the heart, brain, and lungs. This practice supports a smoother transition from intrauterine to extrauterine life, promotes the conversion of respiratory circulation, and can reduce preterm infant mortality by 30%. Additionally, DCC decreases the incidence of complications such as intraventricular hemorrhage, necrotizing enterocolitis, and late-onset sepsis. It also increases blood volume, minimizes the need for blood transfusions, enhances iron storage, and lowers the risk of long-term neurodevelopmental issues. Therefore, DCC emerges as a viable strategy to enhance the perinatal prognosis of preterm infants[4-8]. However, there are limited reports in China regarding the implementation of DCC in premature infants born at less than 30 weeks gestation. The investigators hospital began adopting DCC for preterm infants in 2023 and has developed and standardized the operational procedures for this practice. However, relevant clinical studies have yet to be conducted.

Neonatal respiratory distress syndrome (NRDS) is a condition resulting from a deficiency of pulmonary surfactant (PS) in the alveoli. It is the most common respiratory issue encountered by very premature infants, who often experience progressively worsening respiratory distress shortly after birth. Treatment for NRDS involves respiratory support and the administration of exogenous PS. Traditionally, this is done through tracheal intubation. However, recent clinical studies have demonstrated that minimally invasive surfactant administration (MISA) offers several advantages over tracheal intubation. MISA effectively reduces the need for invasive mechanical ventilation within the first 72 hours and plays a significant role in lowering the incidence of bronchopulmonary dysplasia (BPD)[9].

With advancements in DCC and MISA technology in NICU settings, these approaches have become the preferred options for very premature infants who are breathing spontaneously at birth. To further assess the safety and effectiveness of DCC combined with MISA in the investigators hospital's NICU for premature infants born at less than 30 weeks gestation, the investigators propose this quality improvement study. The study aims to compare the incidence and prognosis of bronchopulmonary dysplasia (BPD) and other complications before and after the implementation of DCC and MISA in the NICU.

The investigators hospital has been implementing MISA since 2017 and has gained extensive clinical experience in treating NRDS in premature infants using this method. The investigators previously conducted a prospective multicenter study comparing MISA with tracheal intubation for surfactant administration shortly after birth. The results indicated that the incidence of bronchopulmonary dysplasia (BPD) and hemodynamically significant patent ductus arteriosus (hsPDA) was lower in the MISA group, highlighting its suitability for premature infants born at less than 30 weeks gestation[10-11]. The investigators hospital has gradually implemented DCC for premature infants prior to this research and has established a comprehensive protocol for its application in the delivery room and during surgical procedures. As a result, the investigators NICU is well-equipped to perform DCC combined with MISA for infants born at less than 30 weeks gestation. Based on previous research findings, this study specifically targets premature infants under 30 weeks, a group that exhibits a relatively high incidence of bronchopulmonary dysplasia (BPD). By monitoring the respiratory and overall health outcomes of these infants following the application of DCC combined with MISA, the investigators aim to evaluate the effectiveness of this NICU quality improvement measure in enhancing the prognosis of very premature infants.

ELIGIBILITY:
Inclusion Criteria ① Infants of 23 to 29+6 weeks GA. ② Born in Peking University Third Hospital, having spontaneous breathing after birth; ③ Diagnosed as NRDS; NRDS is defined as progressive dyspnea that occurs after birth, with or without imaging evidence, excluding other causes of dyspnea.

Exclusion criteria

* Premature infants who have received tracheal intubation prior to the use of PS due to resuscitation or other reasons shortly after birth; ② Premature infants with identified or confirmed congenital abnormalities (such as fetal edema, chylothorax, or neuromuscular disease) or severe birth complications (including hemorrhagic shock, air leakage, or early-onset sepsis) that impact respiratory function.; ③ Newborns who discontinue treatment or have incomplete information; ④ Newborns involved in other intervention research studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a single-center ambispective cohort study involving hospitalized preterm infants in the NICU of Peking University Third Hospital from June 1st, 2017, to May 31th, 2025. The subjects from June 1st, 2017, to May 31 th, 2024, were included in the retrospective cohort study, while a prospective cohort study was conducted from June 1st , 2024, to May 31th, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 518 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
incidence of bronchopulmonary dysplasia | At 36 weeks PMA
  The primary outcome is the incidence of bronchopulmonary dysplasia (BPD) at a corrected gestational age of 36 weeks.

SECONDARY OUTCOMES:
Rate of patent ductus arteriosus with hemodynamic changes | From enrollment to 30 days after birth
  Rate of patent ductus arteriosus with hemodynamic changes
Rate of air leakage, pulmonary hemorrhage, infectious pneumonia | Through study completion and up to corrected three months
  Rate of air leakage, pulmonary hemorrhage, infectious pneumonia
Rate of late onset sepsis with positive blood culture | Through study completion and up to corrected three months
  Rate of late onset sepsis with positive blood culture
Rate of retinopathy of prematurity | Through study completion and up to corrected three months
  Rate of retinopathy of prematurity onset before correcting gestational age for 50 weeks
Rate of III-IV ° periventricular intraventricular hemorrhage and periventricular leukomalacia | Through study completion and up to corrected three months
  Rate of III-IV ° periventricular intraventricular hemorrhage and periventricular leukomalacia
Rate of neonatal necrotizing enterocolitis IIa or above | Through study completion and up to corrected three months
  Rate of neonatal necrotizing enterocolitis IIa or above
Length of hospital stay | From enrollment to the end of treatment at an average of 8 weeks
  Length of hospital stay
In-hospital mortality | Through study completion and up to corrected three months
  In-hospital mortality
Rate of hyperbilirubinemia | Through study completion and up to corrected three months
  Rate of hyperbilirubinemia
First time of blood transfusion during hospitalization | Through study completion and up to corrected three months
  First time of blood transfusion during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Fogarty M, Osborn DA, Askie L, Seidler AL, Hunter K, Lui K, Simes J, Tarnow-Mordi W. Delayed vs early umbilical cord clamping for preterm infants: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Jan;218(1):1-18. doi: 10.1016/j.ajog.2017.10.231. Epub 2017 Oct 30. PMID 29097178
- [Background] Garcia C, Prieto MT, Escudero F, Bosh-Gimenez V, Quesada L, Lewanczyk M, Pertegal M, Delgado JL, Blanco-Carnero JE, De Paco Matallana C. The impact of early versus delayed cord clamping on hematological and cardiovascular changes in preterm newborns between 24 and 34 weeks' gestation: a randomized clinical trial. Arch Gynecol Obstet. 2024 Jun;309(6):2483-2490. doi: 10.1007/s00404-023-07119-0. Epub 2023 Jul 12. PMID 37436461
- [Background] Yoon S, Jin Y, Kim Y, Sung JH, Choi SJ, Oh SY, Roh CR. Effect of delayed cord clamping on maternal and neonatal outcome in twin pregnancies: a retrospective cohort study. Sci Rep. 2023 Oct 13;13(1):17339. doi: 10.1038/s41598-023-44575-9. PMID 37833351
- [Background] McDonald SD. Deferred cord clamping and cord milking: Certainty and quality of the evidence in meta-analyses, and systematic reviews of randomized control trials, guidelines, and implementation studies. Semin Perinatol. 2023 Aug;47(5):151790. doi: 10.1016/j.semperi.2023.151790. Epub 2023 Jun 13. PMID 37349189
- [Background] McDonald SD, Narvey M, Ehman W, Jain V, Cassell K. Guideline No. 424: Umbilical Cord Management in Preterm and Term Infants. J Obstet Gynaecol Can. 2022 Mar;44(3):313-322.e1. doi: 10.1016/j.jogc.2022.01.007. PMID 35300830
- [Background] Jobe AH. Mechanisms of Lung Injury and Bronchopulmonary Dysplasia. Am J Perinatol. 2016 Sep;33(11):1076-8. doi: 10.1055/s-0036-1586107. Epub 2016 Sep 7. PMID 27603539
- [Background] Doyle LW, Carse E, Adams AM, Ranganathan S, Opie G, Cheong JLY; Victorian Infant Collaborative Study Group. Ventilation in Extremely Preterm Infants and Respiratory Function at 8 Years. N Engl J Med. 2017 Jul 27;377(4):329-337. doi: 10.1056/NEJMoa1700827. PMID 28745986
- [Background] Lui K, Lee SK, Kusuda S, Adams M, Vento M, Reichman B, Darlow BA, Lehtonen L, Modi N, Norman M, Hakansson S, Bassler D, Rusconi F, Lodha A, Yang J, Shah PS; International Network for Evaluation of Outcomes (iNeo) of neonates Investigators. Trends in Outcomes for Neonates Born Very Preterm and Very Low Birth Weight in 11 High-Income Countries. J Pediatr. 2019 Dec;215:32-40.e14. doi: 10.1016/j.jpeds.2019.08.020. Epub 2019 Oct 3. PMID 31587861
- [Derived] Zhang Y, Zhang H, Zhang Y, Li X, Yan Z, Zhang J, Zhang H, Piao M, Han T. Impact of delayed cord clamping and minimally invasive surfactant administration on outcomes in premature infants with neonatal respiratory distress syndrome at less than 30 weeks gestation: a NICU quality improvement study. Front Pediatr. 2025 Nov 18;13:1686362. doi: 10.3389/fped.2025.1686362. eCollection 2025. PMID 41341102